CLINICAL TRIAL: NCT04131712
Title: Mechanisms Underlying Local and Systemic Effects of Massage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esther Dupont-Versteegden (Other)
Collaborators: University of Oklahoma (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Esther Dupont-Versteegden, Ph.D., University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 43499; R21AT010847 (NIH)
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Muscle Atrophy
Keywords: Massage; Muscle; Extracellular Vesicles; Atrophy
MeSH Terms: conditions — Muscular Atrophy; Atrophy | interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Primary outcome assessors are blinded to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ambulatory Control (No Intervention): Following baseline assessments, participants will be randomized into the ambulatory group for the remainder of the study. Atrophy will not be induced and massage intervention will not be applied. Ambulatory groups will be recruited following the immobilized groups.
- Ambulatory Massage (Sham Comparator): Following baseline assessments, participants will be randomized into the ambulatory group for the remainder of the study. No atrophy induction. Four massage treatments will be applied every other day until the end of the study. Ambulatory groups will be recruited following the immobilized groups.
  Interventions: Other: Massage
- Immobilization Control (No Intervention): Following baseline assessments, participants will be randomized into the unilateral lower limb suspension group undergoing atrophy for the remainder of the study. Massage intervention will not be applied.
- Immobilization Massage (Experimental): Following baseline assessments, participants will be randomized into the unilateral lower limb suspension group undergoing atrophy for the remainder of the study. Four massage treatments will be applied every other day until the end of the study.
  Interventions: Other: Massage

INTERVENTIONS:
Other: Massage — A custom-made cyclic compressive loading (CCL) device will be used to apply a mechanical load to the left thigh of the participants. Massage application using a 35 Newton load will be applied for 15 minutes every other day over the course of 7 days for a total of four massages.
  Arms: Ambulatory Massage; Immobilization Massage

SUMMARY:
The purpose of this study is to determine whether massage can attenuate the loss of muscle mass in humans after a short period of disuse.

DETAILED DESCRIPTION:
The loss of skeletal muscle mass is a common symptom associated with diseases such as cancer, AIDS, diabetes, and congestive heart failure, and with aging. Muscle atrophy is associated with poor disease prognosis and decreased quality of life and therefore, maintaining muscle size and reducing the loss of muscle during disuse atrophy is of vital significance. Mechanical stimulation of muscle, such as during resistance exercise, stimulates protein synthesis that increases muscle protein content, and muscle size. The investigators have shown that mechanical stimulation applied to skeletal muscle in the form of massage is an effective mechanotherapy in rats, since it leads to a shift in protein turnover favoring anabolism, attenuation of muscle loss and enhanced regrowth after disuse-induced atrophy. Whether the same positive effect of massage occurs in humans is currently unknown, but would be extremely beneficial for skeletal muscle and overall health in case where resistance exercise is contraindicated or not feasible. In addition to the direct anabolic effects on the massaged rat muscle, the investigators have shown an equally beneficial response on the homologous muscle in the contralateral non-massaged limb. This novel finding indicated the existence of indirect mechanisms that could have profound systemic effects beyond the massaged muscle. Extracellular vesicles (EVs) are lipid membrane-bound vesicles released from cells with the ability to modulate function of cells from which they are released, as well as in cells with which they fuse. As such EVs are likely mediators of the well-documented but poorly-understood effects of massage in humans on the brain and other organs, such as relief of pain, anxiety or depression or changes in immunity. Therefore, the goal of this proposal is to determine anabolic effects of massage in human muscle, and to identify whether EVs released with massage are candidates for beneficial effects of this mechanotherapy on muscle as well as other organs. In Aim 1 the investigators will address the following hypothesis: Massage acts as a mechanotherapy by attenuating muscle atrophy through a shift in protein biogenesis towards anabolism in humans. Using a novel massage device we will apply mechanical load to muscle undergoing atrophy through unilateral lower limb suspension and muscle size as well as protein synthesis and degradation will be determined. In Aim 2 the investigators will test the hypothesis that massage attenuates the loss of EVs during atrophy by enhancing EV biogenesis in muscle. The investigators will measure EVs and their miRNA cargo in the serum, and markers of EV biogenesis in muscle of human subjects from Aim 1. Results from this study will indicate not only whether mechanotherapy, such as massage, can attenuate atrophy and enhance anabolic processes during disuse, but also determine whether EVs are a candidate mechanism for the overall health benefits of massage.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-30 years of age.
* All races and ethnic backgrounds.
* Non-smoker and generally healthy.

Exclusion Criteria:

* Have a current lower extremity musculoskeletal injury or compromised musculoskeletal function that would not allow the safe use of crutches or a brace.
* Previous lower extremity surgeries or injury.
* Activities of daily living require long periods of standing or driving a manual transmission car.
* Body mass index (BMI) under 27.
* Evidence or signs and symptoms of metabolic syndrome or disorder (diagnosis of diabetes or insulin resistance, elevated BP, high fasting blood sugar, abnormal cholesterol or triglyceride levels).
* Thyroid disorder.
* Acute or chronic infections.
* Use of systemic steroids, anabolic steroids, or growth hormone.
* Chronic aspirin or NSAID use (unless it can be safely stopped prior to the biopsies), and any other use of an anticoagulant (e.g., Coumadin) or history of bleeding including history of hypo- or hyper-coagulation disorders.
* Lidocaine allergy (1% lidocaine is the local anesthetic used during the muscle biopsy procedure).
* Any other condition or events considered exclusionary by the PI and/or physician, such as non-compliance.
* Pregnancy.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Dupont-Versteegden, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were actively recruited from the University of Kentucky campus as well as from the surrounding Lexington community through local advertisement using IRB approved recruitment flyers or newspaper advertisement. Recruitment occurred between August of 2020 and May 2023.
  The COVID pandemic shut down research activities at the University of Kentucky for some time impacting recruitment. Thus, the PI decided to focus on randomization of immobilized groups
Pre-assignment Details: Consent, inclusion/exclusion criteria checklist, participant characteristics such as height and weight, and pregnancy testing were conducted prior to randomization.
Period: Overall Study
Arm/Group | Ambulatory Control | Ambulatory Massage | Immobilization Control | Immobilization Massage
Started | 9 | 0 | 19 | 16
Completed | 9 | 0 | 16 | 16
Not Completed | 0 | 0 | 3 | 0
Not completed — COVID related | 0 | 0 | 2 | 0
Not completed — PI withdrawal, subject could not follow study schedule | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: More focus was placed on immobilization groups during COVID. The ambulatory massage group was not recruited as a result.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambulatory Control | Ambulatory Massage | Immobilization Control | Immobilization Massage | Total
Number analyzed (Participants) | 9 | 0 | 16 | 16 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0 | 0 | 0
  Between 18 and 65 years | 9 |  | 16 | 16 | 41
  >=65 years | 0 |  | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.83 (3.31) |  | 22.64 (3.93) | 22.07 (3.77) | 22.46 (3.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  | 12 | 12 | 28
  Male | 5 |  | 4 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 1 | 3 | 5
  Not Hispanic or Latino | 8 |  | 15 | 13 | 36
  Unknown or Not Reported | 0 |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0 | 0
  Asian | 1 |  | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0 | 0
  Black or African American | 0 |  | 1 | 2 | 3
  White | 8 |  | 15 | 14 | 37
  More than one race | 0 |  | 0 | 0 | 0
  Unknown or Not Reported | 0 |  | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 |  | 16 | 16 | 41

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Myofiber Cross Sectional Area (CSA).
Description: The ability of massage to attenuate the atrophic response to disuse will be determined. Muscle biopsies of the vastus lateralis will be used to quantify myofiber cross-sectional area. The percent change in myofiber size between day 7 and day -2 was used.
  Calculation details: [(day 7 CSA) - (day -2 CSA)/(day -2 CSA)]*100
Time Frame: 9 days
Population: Only one biopsy post 9 days was taken in the ambulatory groups only and thus % change could not be calculated. For the immobilization control group, one biopsy specimen could not be accurately analyzed due to tissue quality.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Ambulatory Control | Ambulatory Massage | Immobilization Control | Immobilization Massage
Number analyzed (Participants) | 0 | 0 | 15 | 16
percent change from baseline |  |  | -15.1 (5.1) | -13.4 (3.0)

2. Primary Outcome: Myofibrillar Protein Synthesis Rate (MyoKsyn).
Description: The ability of massage to attenuate the atrophic response to disuse due to protein synthesis will be determined. Muscle biopsies of the vastus lateralis will be used to quantify protein synthesis rates.
Time Frame: 9 days
Population: Participants were not randomized to the ambulatory massage group. For the immobilization control group, one biopsy specimen could not be accurately analyzed due to tissue quality.
Measure: Mean (Standard Deviation); unit: percentage of protein produced per day
Arm/Group | Ambulatory Control | Ambulatory Massage | Immobilization Control | Immobilization Massage
Number analyzed (Participants) | 8 | 0 | 15 | 16
percentage of protein produced per day | 1.19 (0.25) |  | 1.04 (0.31) | 1.07 (0.29)

3. Secondary Outcome: Percent Change in Serum Extracellular Vesicle Number (EV #).
Description: The ability of massage to attenuate the loss in EV number will be determined. Serum will be used to quantify EV numbers. The percent change in EVs between day 7 and day -2 was used.
Time Frame: 9 days
Population: Data was not generated.
Arm/Group | Ambulatory Control | Ambulatory Massage | Immobilization Control | Immobilization Massage
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Percent Change in the Expression of Muscle Rab27b mRNA.
Description: The ability of massage to attenuate the loss in Rab27b protein expression will be determined. Muscle biopsies of the vastus lateralis will be used to quantify muscle Rab27b expression. The percent change in muscle Rab27b expression between day 7 and day -2 was used.
Time Frame: 9 days
Population: Data was not generated.
Arm/Group | Ambulatory Control | Ambulatory Massage | Immobilization Control | Immobilization Massage
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over the 9 day study period and for approximately 3 days post last biopsy.
Description: AEs and SAEs were collected according to the standard definitions used by clinicaltrials.gov.
Arm/Group | Ambulatory Control | Ambulatory Massage | Immobilization Control | Immobilization Massage
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/0 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/0 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/9 | 0/0 | 4/16 | 5/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambulatory Control (N=9) | Ambulatory Massage (N=0) | Immobilization Control (N=16) | Immobilization Massage (N=16)
Nausea (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Persistent pain following biopsy
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) — Blister forming underneath steri-strip applied following bioppsy.
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Participant reported feeling more fatigue after ingesting heavy water

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT04131712/Prot_002.pdf
  • Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT04131712/SAP_003.pdf
  • Informed Consent Form (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT04131712/ICF_001.pdf